CLINICAL TRIAL: NCT07122531
Title: Metabolic and Clinical Evaluation of Medium-Chain Triglyceride-Based Exogenous Ketone Supplementation as an Adjunctive Treatment for First-Episode Psychosis
Brief Title: Recovery With Exogenous Ketones and Antipsychotics
Acronym: RECAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Stephen Cunnane, Professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025 -5840
Record Dates: First submitted 2025-08-05; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: First Episode Psychosis
Keywords: first episode psychosis; Schizophrenia; metabolism; ketone; medium triglyceride; antipsychosis; glucose
MeSH Terms: conditions — Schizophrenia; Ketosis

STUDY DESIGN:
Intervention Model Description: Uncontrolled prospective pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12 week ketogenic supplementation (Experimental): Supplementation with 15 g of medium chain triglyceride oil, emulsified in beverage of choice, twice daily (morning and evening) for 12 weeks,.
  Interventions: Other: Medium chain triglyceride oil

INTERVENTIONS:
Other: Medium chain triglyceride oil — Supplementation with 15 g of medium chain triglyceride oil, a food product commercially available over-the-counter in regular grocery stores, emulsified in beverage of choice, twice daily (morning and evening) for 12 weeks.

SUMMARY:
The RECAP project will evaluate the clinical and metabolic effects of adding exogenous ketones to antipsychotic (AP) treatment in young adults with a first episode of psychosis (FEP).

FEP requires early intervention to limit relapse, chronic symptoms, cognitive decline, and reduced life expectancy. Symptoms include positive (hallucinations, delusions), negative (amotivation, anhedonia), cognitive (attention, working memory), and mood disturbances. Standard care combines second- or third-generation APs with psychosocial interventions. However, many patients have persistent symptoms despite optimal treatment.

Psychosis is linked to increased cardiovascular and obesity risk. APs can cause insulin resistance, type 2 diabetes, and dyslipidemia, but some metabolic abnormalities-both systemic and cerebral-may precede AP use, suggesting an intrinsic metabolic dysfunction. Brain energy metabolism is often impaired, with altered insulin signaling, glucose transport, and ATP production. Glucose hypometabolism in the prefrontal cortex correlates with negative and cognitive symptoms, even before medication, resembling patterns in Alzheimer's, bipolar disorder, and depression.

Ketones, especially beta-hydroxybutyrate, provide an alternative to glucose for brain energy. Ketogenic diets have therapeutic potential but are difficult to maintain, particularly in psychiatric populations. Exogenous ketones, such as medium-chain triglycerides (MCTs), can raise circulating ketone levels without major dietary changes. MCT supplementation has been shown to improve brain metabolism and cognition in other conditions, but no studies have tested it in FEP.

This uncontrolled, prospective pilot study will provide 15 g of MCT oil twice daily for 12 weeks, in addition to participants' usual diet and treatment. The primary objective is to assess changes in circulating ketone levels and metabolic markers (glucose, insulin, HbA1c). Secondary objectives include feasibility, acceptability, effects on real-time glucose metabolism (via continuous glucose monitoring), clinical symptoms (negative, cognitive), quality of life, other metabolic biomarkers, and general systemic markers.

This is the first study to test exogenous ketones in FEP. It will assess safety, tolerability, and potential metabolic and clinical benefits, offering preliminary mechanistic insights and guiding future integrative mental health strategies.

ELIGIBILITY:
Inclusion Criteria:

* Referred or self-referred to the PEP Clinic of the Estrie region, either as an outpatient or inpatient.
* Currently receiving a second- or third-generation antipsychotic at a stable dose for at least 4 weeks.
* Able to read and communicate in French or English.
* Capable of understanding and signing the informed consent form.

Exclusion Criteria:

* Pregnancy, childbirth within the past 6 months, or breastfeeding.
* any use of MCT oil, ketone salts, or a ketogenic diet within the past year.
* Previous diagnosis of type I or type II diabetes.
* Uncontrolled acute suicidal ideation at the time of inclusion in the PEP clinic.
* Other conditions that may interfere with participation, as determined by the qualified physician.
* Pancreatitis (inflammation of the pancreas) or liver failure.
* Metabolic condition affecting fat metabolism or inherited carnitine deficiency and its related enzymes.
* Porphyria.
* Pyruvate kinase deficiency.
* Neurodevelopmental disorder of unknown etiology or rare genetic disease.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Plasma total ketones concentration | 12 weeks
  Change in plasma total ketone (acetoacetate + betahydroxybutyrate) after 12 weeks of supplementation (uM)
Plasmatic glucose concentration | 12 weeks
  Change in glucose concentration (mM) after 12 weeks of supplementation (uM)
Plasma Insulin concentraiton | 12 weeks
  Change in insuline concentration (UI) after 12 weeks of supplementation (uM)
Plasma Glycated hemoglobin | 12 weeks
  Change in Glycated hemoglobin (%) after 12 weeks of supplementation

SECONDARY OUTCOMES:
acceptability of exogenous ketone supplementation | at the end of the 12 weeks treatment
  Participant perspectives will be collected through a short semi-structured interview and analyzed using a descriptive thematic approach.
compliance rate | during 12 weeks intervention
  dose of supplement taken during the 12 weeks/ number of dose expected (%)
Adverse event rate | 12 weeks intervention
  Total number of adverse event during the intervention
Drop-out rate | After 12 weeks of intervention
  Number of participant taht have drop-out/total number of participant included in the study
Glucose average (mean of glucose measured by continuous glucose monitoring) | 12 weeks
  Change in mean plasma glucose concentration (mM) measured by continuous glucose monitoring (CGM) over the course of 8 days; after 12 weeks intervention.
glucose variability (SD of glucose measured by continuous glucose monitoring) | 12 weeks
  coefficient of variation of plasma glucose concentration (%) measured by systemic glucose metabolism using continuous glucose monitoring (CGM) over the course of 8 days.
Negative symptomes | 12 weeks
  Change in the score of the Scale for the assessment of negative symptoms (SANS) (score 0 to 125 with worsening of symptom with higher result)
Depression status measured by the score of "Calgary Depression Scale for Schizophrenia | 12 weeks
  Change int Score of "Calgary Depression Scale for Schizophrenia" (CDSS) . Min score 0, maximum score 27 with worsening of the patient condition with hight value
Brief Assessment of Cognition (BACS) | 12 weeks
  Change in composite score (express as Z score) of the brief assessment of cogition
Functionning level measured by the score of the Global Assessment of functionning | 12 weeks
  Change in the Score of the "Global Assessment of functionning (GAF). Min score 0, maximum score 100, with worsening of the patient condition with higher value

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Zemmour, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Hotel-Dieu CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No